CLINICAL TRIAL: NCT01132079
Title: Role for Pimecrolimus in Restoring Skin Barrier Function and Normalizing Epidermal Lipid Content and Differentiation in Atopic Epidermis: a Randomized, Intra-patient, Double-blind (Right/Left Arm) Study in Adults With Atopic Dermatitis Treated With 1 % Pimecrolimus Cream and 0.1 % Betamethasone Cream as Treatment Control Twice Daily for 3 Weeks
Brief Title: Pimecrolimus and Epidermal Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: Deutsche Forschungsgemeinschaft, Bonn, Germany (Unknown); Novartis Pharma GmbH, Nürnberg, Germany (Unknown)
Responsible Party: Ehrhardt Proksch, MD, PhD, Dept. of Dermatology, Venerology and Allergology, University Hospitals of Schleswig-Holstein, Campus Kiel, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Protocol No. ELBE-2005
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2005-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; barrier function; pimecrolimus
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pimecrolimus cream treatment (Experimental)
  Interventions: Drug: cream treatment
- Betamethasone valerate cream treatment (Active Comparator)
  Interventions: Drug: cream treatment

INTERVENTIONS:
Drug: cream treatment

SUMMARY:
This study seeks to investigate the role of pimecrolimus in restoring disturbed skin barrier function and reversing epidermal abnormalities found in atopic dermatitis (AD). The project is based on findings the investigators presented at the recent SID meeting in Providence and published in the J Invest Dermatol (122: 1423-31, 2004). The investigators research shows that AD is characterized by impaired skin barrier function, reduced stratum corneum hydration, impaired epidermal lipid composition and epidermal differentiation. In this proposed project, the investigators wish to examine the influence of pimecrolimus and betamethasone valerate on transepidermal water loss (TEWL) as a marker of the skin barrier function, on stratum corneum hydration, on stratum corneum lipid content and on epidermal differentiation regarding keratins and cornified envelope proteins in AD patients. The study involves biophysical measurements of TEWL and skin hydration, lipid analysis, immuno-histochemistry, Western blotting and micro array techniques. This study shall clarify whether pimecrolimus restores the epidermal barrier and whether this contributes to the beneficial effect of pimecrolimus on AD.

Objectives:

To explore the stratum corneum hydration, transepidermal water loss, capacity for barrier repair and the integrity of the stratum corneum in patients treated with 1 % pimecrolimus cream when applied twice a day to atopic dermatitis of the upper limbs, and to access the substance's influences on the epidermis through histological, ultra-structural, and biochemical analysis using punch biopsies from day 1 of one arm and day 22 from both treated arms. 0.1 % betamethasone valerate cream b.i.d will be used as a control treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included only if the following apply at the baseline visit (day 0, before first application of study medication).

Patients to be included are:

* Males and females of any race.
* >= 18 years old.
* Have atopic dermatitis as defined by Hanifin and Rajka criteria.
* History of mild to moderate atopic dermatitis
* At least 10 % of each upper limb affected by atopic dermatitis excluding the surface area of the hands, as these will not be treated in order to avoid cross-contamination. As reference: one hand (palm and fingers) corresponds to 10% of patient's upper limb surface.
* One specific, representative area of the disease on each upper limb with similar size and severity on both upper limbs. These will be considered the target lesions.
* A target lesion score of at least 3 to 8 (on a scale of 0-12) for both right and left target lesions and not differing more than 1 score point between the right and left sides.
* be able to suspended treatment of atopic dermatitis with other therapies for the duration of the study (4-6 weeks).
* Must be informed of study procedures and have signed the informed consent form approved for the study.

Exclusion Criteria:

Females:

* Who are pregnant or breastfeeding.
* Who are menstruating, capable of becoming pregnant and not practicing a medically approved method of contraception. "Medically approved" contraceptive may, at the discretion of the investigator, include abstinence. (If patients are on oral contraceptives, they must have begun treatment at least one month prior to baseline and continue at least four weeks after the last treatment).

Other therapies/medications:

* Prior phototherapy or systemic therapy known to or suspected to have an effect on atopic dermatitis within 14 days prior to first application of study medication. Patients on a low stable dose of inhaled steroids (dose known to have negligible systemic absorption) and systemic antihistamines may participate.
* Topical therapy known to or suspected to have an effect on atopic dermatitis (including topical steroids, topical tacrolimus ointment or topical pimecrolimus cream) on the upper limbs within 7 days prior to first application of study medication.
* Topical therapy known to or suspected to have an effect on atopic dermatitis on other areas than upper limbs if total body surface treated is higher than 20% (due to the higher risk of systemic absorption affecting the lesions of the upper limbs) within 7 days prior to first application of study medication

Concurrent diseases / conditions and history of their diseases / conditions:

* Patients who have signs of skin atrophy and corticoid damage on the target areas
* Patients who are immunocompromised (e.g. lymphoma, AIDS, Wiskott-Aldrich Syndrome)
* Patients who have concurrent skin disease (e.g. impetigo) on or near the study area which could interfere with study evaluations
* Patients who have acute viral skin infections (e.g. herpes simplex, varicella zoster) Investigational drug / therapy use.
* Patients who have used investigational drugs within 8 weeks prior to first application of study medication or intend to use other investigational drugs during the course of the study Ingredient hypersensitivity
* Patients with known hypersensitivity to any ingredient of the study medication (see technical information sheet) Compliance / reliability / investigator judgment
* Patients who who are, in the opinion of the investigator, known to be unreliable or non-compliant with medical treatment, or are known to miss appointments (according to patient records)
* Patients who drug abuse problems, mental dysfunction or other factors limiting their ability to cooperate fully
* Patients who any other condition or prior/present treatment which, in the opinion of the investigator, will render the patient ineligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03

PRIMARY OUTCOMES:
To explore the effect of 1 % pimecrolimus cream on the epidermis in adults with AD
  To explore the effect of 1 % pimecrolimus cream on the epidermis in adults with AD (with 0.1 % betamethasone serving as control) by testing the hypothesis that:
  1. 1 % pimecrolimus cream leads to a reduction of biophysical parameters of AD representing the permeability barrier of the skin after three weeks of treatment.
  2. To explore the epidermal effect on proliferation rate, differentiation, and stratum corneum lipid content.

SECONDARY OUTCOMES:
To explore the effect of 1 % pimecrolimus cream induced changes in ultra-structure and gene expression in the epidermis
  1. To explore the effect of 1 % pimecrolimus cream induced changes in ultra-structure and gene expression in the epidermis.
  2. To compare the key protein molecules of keratinocyte growth and differentiation and their gene expression in relationship to clinical skin improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ehrhardt Proksch, MD, PhD, Principal Investigator — Dept. of Dermatology, University of Kiel
Locations (1):
- Dept. of Dermatology, University of Kiel, Kiel, Germany

REFERENCES:
- [Result] Jensen JM, Pfeiffer S, Witt M, Brautigam M, Neumann C, Weichenthal M, Schwarz T, Folster-Holst R, Proksch E. Different effects of pimecrolimus and betamethasone on the skin barrier in patients with atopic dermatitis. J Allergy Clin Immunol. 2009 May;123(5):1124-33. doi: 10.1016/j.jaci.2009.03.032. PMID 19410693
- [Result] Jensen JM, Pfeiffer S, Witt M, Brautigam M, Neumann C, Weichenthal M, Schwarz T, Folster-Holst R, Proksch E. Different effects of pimecrolimus and betamethasone on the skin barrier in patients with atopic dermatitis. J Allergy Clin Immunol. 2009 Sep;124(3 Suppl 2):R19-28. doi: 10.1016/j.jaci.2009.07.015. PMID 19720208